CLINICAL TRIAL: NCT04758468
Title: Effects of Telerehabilitation-Based Pelvic Floor Muscle Training on Urinary Incontinence, Sexual Function and Quality of Life in People With Multiple Sclerosis
Brief Title: Effects of Telerehabilitation-Based Pelvic Floor Muscle Training in People With Multiple Sclerosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dokuz Eylul University (Other)
Collaborators: Izmir Katip Celebi University (Other)
Responsible Party: Principal Investigator, Turhan Kahraman, Associate Professor, Dokuz Eylul University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 5742-GOA
Record Dates: First submitted 2021-02-11; First posted 2021-02-17 (Actual); Last update posted 2022-03-29 (Actual); Status verified 2022-03

CONDITIONS: Multiple Sclerosis; Urinary Incontinence
Keywords: Multiple Sclerosis; Urinary Incontinence; Pelvic Floor Muscle Training; Sexual Function
MeSH Terms: conditions — Multiple Sclerosis; Urinary Incontinence

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Telerehabilitation-based pelvic floor muscle training (Experimental)
  Interventions: Behavioral: Telerehabilitation-based pelvic floor muscle training
- Home-based pelvic floor muscle training (Active Comparator)
  Interventions: Behavioral: Home-based pelvic floor muscle training
- Control (no specific intervention) (No Intervention)

INTERVENTIONS:
Behavioral: Telerehabilitation-based pelvic floor muscle training — Telerehabilitation-based pelvic floor muscle training group will individually receive telerehabilitation-based pelvic floor muscle training under the guidance of a physiotherapist 2 sessions per week for 8 weeks. Participants will do their exercises themselves 2 times on the days where sessions are held with a physiotherapist. Participants will continue to exercise 3 times a day in the remaining days.
  Both intervention groups will follow the same pelvic floor muscle training protocol for 8 weeks.
  Arms: Telerehabilitation-based pelvic floor muscle training
Behavioral: Home-based pelvic floor muscle training — The home-based pelvic floor muscle training group will do their individual exercises 3 times a day for 8 weeks.
  Both intervention groups will follow the same pelvic floor muscle training protocol for 8 weeks.
  Arms: Home-based pelvic floor muscle training

SUMMARY:
The effectiveness of pelvic floor muscle training on urinary incontinence and sexual function has been known for many years. However, the evaluation of its effectiveness in people with Multiple Sclerosis (MS) has recently begun and the level of evidence is limited. In addition, the applicability of pelvic floor muscle training based on telerehabilitation in the presence of a physiotherapist has not been investigated before.

The aims of this study;

1. The main aim of this study is to evaluate the feasibility and acceptability of telerehabilitation-based pelvic floor muscle training under the guidance of a physiotherapist, which will be applied for the first time.
2. Another aim is to compare this method with the effects of not receiving treatment other than usual treatment or receiving home-based pelvic floor muscle training on urinary incontinence, sexual dysfunction and psychosocial outcomes.

The participants will randomly be allocated into three groups: (1) Telerehabilitation-based pelvic floor muscle training, (2) Home-based pelvic floor muscle training, and (3) Control group Telerehabilitation-based pelvic floor muscle training group will individually receive telerehabilitation-based pelvic floor muscle training under the guidance of a physiotherapist 2 sessions per week for 8 weeks. Participants will do their exercises themselves 2 times on the days where sessions are held with a physiotherapist. Participants will continue to exercise 3 times a day in the remaining days. The home-based pelvic floor muscle training group will do their individual exercises 3 times a day for 8 weeks. The control group will receive no specific training

DETAILED DESCRIPTION:
Both intervention groups will follow the same pelvic floor muscle training protocol for 8 weeks, but the home-based group will follow the exercise protocol individually while the telerehabilitation-based group will follow the telerehabilitation-based under the guidance of the physiotherapist.

Exercises will be applied 3 times a day according to the specified protocol. An information leaflet will be distributed to the home exercise group. The telerehabilitation-based group will receive telerehabilitation-based pelvic floor muscle training under the guidance of a physiotherapist individually for 2 sessions a week, the patient will do the exercises twice a day in the days of the sessions with the physiotherapist, and the remaining days will continue to do it 3 times a day like a home exercise group. The control group will not receive treatment other than their routine treatment, and the patients will be informed that they will be treated if they wish at the end of the study.

The progression in Pelvic Floor Muscle Training will be achieved by increasing the exercise volume and diversifying the positions. The assessments will be applied at baseline, 4, 8, and 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Having been diagnosed with MS according to McDonald diagnostic criteria
* Having urinary incontinence
* EDSS score less than 8
* Have the cognitive capacity to complete the assessment and treatment protocol

Exclusion Criteria:

* Pregnancy
* Pelvic surgery history
* A history of cesarean or vaginal delivery within 6 months prior to the study
* Progressive disability (1 point increase in EDSS) or attacks in the last 3 months
* Having received pelvic floor muscle training in the last 6 months
* Have had or are receiving treatment for pelvic organ prolapse Patients receiving pharmacological therapy for incontinence whose dose has not changed over the past 3 months will be included, but will be excluded if the dose changes during the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2021-02-18 (Actual); Primary Completion 2021-11-15 (Actual); Study Completion 2021-11-15 (Actual)

PRIMARY OUTCOMES:
Feasibility of the methods-minimum recruitment rate | Through Study Completion, an Average of 8 Weeks
  A minimum recruitment rate of 10 participants per month will be accepted as feasible.
Feasibility of the methods-minimum retention rate | Through Study Completion, an Average of 8 Weeks
  A target retention rate of 80% will be accepted as feasible.
Feasibility of the methods-minimum adherence rate | Through Study Completion, an Average of 8 Weeks
  A target minimum adherence rate of 70% of the overall practice sessions will be accepted as feasible.
Feasibility of the methods-adverse events | Through Study Completion, an Average of 8 Weeks
  A record sheet was prepared for possible adverse events during the tests and intervention. It includes information about seriousness, expectedness, severity, causality, time, duration of the event and clinical action taken. The numbers of adverse events will be reported.
Change in Leakage Episodes | The assessments will be applied at baseline, 4, 8, and 12 weeks.
  The bladder diary is a form that is used to objectively evaluate the frequency and severity of urinary incontinence. It will be used to determine the leakage episodes. It will be filled in three days by the patients. The amount of fluid taken in the diary, the amount of urine, the number of incontinence and pad change are recorded.

SECONDARY OUTCOMES:
Expanded Disability Status Scale (EDSS) | The assessment will be applied at baseline.
  EDSS is the most frequently used scale in evaluating the disability of individuals with MS. Scoring based on neurological examination findings takes a value between 0-10. While 0 shows normal neurological findings, 10 means death due to MS. In this scale in which pyramidal, cerebral, cerebellar, visual, sensory, brainstem, bladder and bowel functions are scored, the best performance of the patient without any special effort is evaluated.
Change in Patient-Determined Disease Steps Scale (PDDS) Score | The assessments will be applied at baseline and 8 weeks.
  PDDS was designed in 1995 as a self-reported outcome measure to enable neurologists without EDSS evaluator certification to measure the level of disability of people with MS. It consists of one question. In PDDS, the patient is asked to choose one of the 9 items that best describes his current walking ability.
Change in Brief International Cognitive Assessment for MS-Symbol Digit Modalities Test Score | The assessments will be applied at baseline and 8 weeks.
  Brief International Cognitive Assessment for MS (BICAMS) has been proposed by an expert panel as a tool for brief cognitive monitoring of individuals with MS in clinical settings.
  Processing speed will be assessed with the Symbol Digit Modalities Test, a subsection of BICAMS.
Change in Brief International Cognitive Assessment for MS-California Verbal Learning Test-Second Edition Score | The assessments will be applied at baseline and 8 weeks.
  Brief International Cognitive Assessment for MS (BICAMS) has been proposed by an expert panel as a tool for brief cognitive monitoring of individuals with MS in clinical settings.
  Verbal learning and memory will be assessed with the California Verbal Learning Test-Second Edition, a subsection of BICAMS.
Change in Brief International Cognitive Assessment for MS-Brief Visuospatial Memory Test-Revised Score | The assessments will be applied at baseline and 8 weeks.
  Brief International Cognitive Assessment for MS (BICAMS) has been proposed by an expert panel as a tool for brief cognitive monitoring of individuals with MS in clinical settings.
  Visual-spatial learning and memory will be assessed with the Brief Visuospatial Memory Test-Revised, a subsection of BICAMS.
Change in Pad Usage | The assessments will be applied at baseline, 4, 8, and 12 weeks.
  The bladder diary is a form that is used to objectively evaluate the frequency and severity of urinary incontinence. It will be used to determine the pad usage. It will be filled in three days by the patients. The amount of fluid taken in the diary, the amount of urine, the number of incontinence and pad change are recorded.
Change in International Consultation on Incontinence Questionnaire-Urinary Incontinence Short Form Score | The assessments will be applied at baseline, 4, 8, and 12 weeks.
  International Consultation on Incontinence Questionnaire-Urinary Incontinence Short Form was developed to evaluate the effect of urinary incontinence and urinary incontinence on quality of life. The scale has four dimensions. The first dimension questions the frequency of urinary incontinence, the second dimension questions the amount of incontinence, the third dimension questions the effect of urinary incontinence on daily life, and the fourth dimension questions the conditions that cause urinary incontinence. In the evaluation, the first three dimensions are scored. Responses to the fourth dimension are used to determine the type of urinary incontinence based on the individual's complaints. The scores that can be obtained from the scale range from 0-21; a low score indicates that urinary incontinence affects the quality of lifeless, while a high score indicates that it affects a lot.
Change in Overactive Bladder-Validated 8-Question (OAB-V8) Score | The assessments will be applied at baseline, 4, 8, and 12 weeks.
  The OAB-V8 is a screening and awareness test that is used to evaluate the symptoms of urgency, urination, frequent urination and feeling of urine at night and waking up in the overactive bladder. The scale consists of 8 items and answers are scored on a 6-level Likert scale. A maximum score of 40 can be obtained from the scale, and a score below 8 eliminates overactive bladder.
Change in EuroQOL 5-Dimension 3-Level Questionnaire Score | The assessments will be applied at baseline, 4, 8, and 12 weeks.
  EuroQOL 5-Dimension 3-Level is a self-report scale developed to evaluate the quality of life and consists of two parts. The first part contains five dimensions. These dimensions are mobility, self-care, usual daily activities, pain/discomfort, and anxiety/depression. These five dimensions are evaluated with one question each. Answers to each dimension; It is scored between 1 and 3. The second part includes a visual analog scale in which the respondents evaluate their current health status between 0 and 100.
Change in Multiple Sclerosis Intimacy and Sexuality Questionnaire-19 (MSISQ-19) Score | The assessments will be applied at baseline, 4, 8, and 12 weeks.
  MSISQ-19 is a test that standardizes primary (direct result of demyelinating lesions), secondary (consequence of other symptoms) and tertiary (related to psychological, emotional, social and cultural factors) sexual dysfunction in the MS population in the last 6 months. It consists of 19 questions and is based on self-assessment in sexual activity and satisfaction. It is scored between 1 and 5.
Change in Hospital Anxiety and Depression Scale (HADS) Score | The assessments will be applied at baseline, 4, 8, and 12 weeks.
  HADS is used to determine the risk of anxiety and depression in the patient and to measure its level and severity. It is a self-report scale consisting of 7 anxiety and 7 depression related questions in total and two subscales. Items are scored with a 3-level Likert-type scale. Higher scores indicate more symptoms.
Change in the number of falls due to a sense of urgency | The assessments will be applied at baseline and 8 weeks.
  The number of falls will be questioned because of the sensing of impingement in the last three months.

CONTACTS AND LOCATIONS:
Locations (1):
- Dokuz Eylul University Hospital, MS Outpatient Clinic, Izmir, Inciralti, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yavas I, Kahraman T, Sagici O, Ozdogar AT, Yigit P, Baba C, Ozakbas S. Feasibility of Telerehabilitation-Based Pelvic Floor Muscle Training for Urinary Incontinence in People With Multiple Sclerosis: A Randomized, Controlled, Assessor-Blinded Study. J Neurol Phys Ther. 2023 Oct 1;47(4):217-226. doi: 10.1097/NPT.0000000000000448. Epub 2023 Jun 12. PMID 37306430